CLINICAL TRIAL: NCT00654121
Title: Prevention of Clinical Onset of Type 1 Diabetes by Daily Administration of Metabolically Active Insulin in High Risk First Degree Relatives.
Brief Title: Prevention of Clinical Onset of Type 1 Diabetes in High Risk First Degree Relatives
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AZ-VUB (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Prof. F Gorus, Free University Brussels
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EVDM IT 001
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2008-04-07 (Estimated); Status verified 2008-04

CONDITIONS: Diabetes, Type I
Keywords: prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 56 subjects will receive metabolically active insulin by subcutaneous injections for 36 months (twice daily)
  Interventions: Drug: Actrapid HM
- 2 (No Intervention)

INTERVENTIONS:
Drug: Actrapid HM — 56 subjects will receive metabolically active insulin by subcutaneous injections for 36 months (twice daily)
  Arms: 1

SUMMARY:
Prophylactic administration of metabolically active insulin can prevent or delay clinical onset of diabetes in a high risk group of nondiabetic siblings as defined by positivity for autoantibodies against IA-2 (IA-2-A).

DETAILED DESCRIPTION:
Hypotheses:

Primary: Prophylactic administration of metabolically active insulin can prevent or delay clinical onset of diabetes in a high risk group of nondiabetic siblings as defined by positivity for autoantibodies against IA-2 (IA-2-A).

Secondary: 1) Untreated siblings with positivity for IA-2-A develop clinical diabetes significantly faster than untreated offspring with the same marker positivity. 2) Plasma proinsulin levels increase disproportionately before clinical onset of Type 1 diabetes both in siblings and offspring. 3) Prophylactic administration of metabolically active insulin reduces the plasma proinsulin/C-peptide ratio in non-diabetic antibody positive siblings and offspring. 4) Prophylactic administration of metabolically active insulin reduces the presence and/or levels of diabetes-associated autoantibodies directed against islet cell components.

Endpoints: Fasting glycemia; fasting and stimulated plasma C-peptide and proinsulin values; islet cell autoantibodies; incidence of hypoglycemia; body weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Sibling/offspring of a Type 1 diabetic patient
* in good general condition
* age 5-39 years
* fasting plasma glucose <126 mg/dL AND an OGTT that is non-diabetic by 1997 ADA criteria (33):

  1. Normal glycemia:

     * fasting plasma glucose < 110 mg/dL and
     * 2 hour plasma glucose < 140 mg/dL
  2. Impaired Fasting Glucose (IFG):

     * fasting plasma glucose 110-125 mg/dL and
     * 2 hour plasma glucose < 140 mg/dL
  3. Impaired Glucose Tolerance (IGT):

     * fasting plasma glucose <110 mg/dL and
     * 2 hour plasma glucose 140-199 mg/dL
* at least positive for IA-2-A
* absence of a protective DQ genotype: A4-B2/X or X/Y or X/X where X = A2-B3.3, A1-B1.9, A1-B1.2, A4-B3.1, A2-B2 or A4.23-B3.1 Y = A1-B1.1, A1-B2, A1-B1.AZH, A3-B2, A3-B3.1, A3-B3.3, A3-B4, A4-B4, A4.23-B4, A4-B3.2, A3-B1.1, A4-B3.3, A4-B1.1 or A4.23-B2 (32)
* cooperative and reliable subject (age ≥ 14 yrs) / parents (age < 14 yrs) giving informed consent by signature; the patient/parents should be informed in sufficient detail on the content and procedure of the protocol, indicating potential risks of insulin therapy; early intervention with metabolically active insulin treatment should be identified as a clinical trial. Both parents should sign and agree with the protocol procedure.

Exclusion Criteria:

* diabetes by 1997 ADA criteria (33):

  * fasting plasma glucose ≥ 126 mg/dL, or
  * 2 hour plasma glucose ≥ 200 mg/dL
* donation of blood during the study or within one month prior to screening
* pregnancy or lactation in women
* use of inadequate anticonception by female patients of childbearing potential
* use of illicit drugs or overconsumption of alcohol (> 3 beers/day) or history of drug or alcohol abuse
* being legally incapacitated, having significant emotional problems at the time of the study, or having a history of psychiatric disorders
* having received antidepressant medications during the last 6 months
* treatment with immune modulating or diabetogenic medication (such as corticosteroids)
* presently participating in another clinical study or having done so during the last 12 months
* history of any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risks to the patient

Ages: 5 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2000-02; Primary Completion 2004-04 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Fasting glycemia; | 2004
fasting and stimulated plasma C-peptide and proinsulin values; | 2004
islet cell autoantibodies; | 2004
body weight gain. | 2004

CONTACTS AND LOCATIONS:
Overall Officials: Frans Gorus, MD,PhD, Principal Investigator — Universitair Ziekenhuis Brussel; Evy Vandemeulebroucke, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (3):
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Academisch Ziekenhuis and Diabetes Research Center - Brussels Free University-VUB, Brussels
  - Department of Endocrinology and Nephrology, UZ Gasthuisberg, Katholieke Universiteit Leuven -KUL, Leuven

REFERENCES:
- [Background] Decochez K, Truyen I, van der Auwera B, Weets I, Vandemeulebroucke E, de Leeuw IH, Keymeulen B, Mathieu C, Rottiers R, Pipeleers DG, Gorus FK; Belgian Diabetes Registry. Combined positivity for HLA DQ2/DQ8 and IA-2 antibodies defines population at high risk of developing type 1 diabetes. Diabetologia. 2005 Apr;48(4):687-94. doi: 10.1007/s00125-005-1702-x. Epub 2005 Mar 9. PMID 15756536
- [Background] Gorus FK, Weets I, Decochez K, van der Auwera BJ. [Preventative biology of type 1 diabetes: implications for clinical preventative studies]. Verh K Acad Geneeskd Belg. 2003;65(4):203-29; discussion 229-31. Dutch. PMID 14534938
- [Background] Decochez K, De Leeuw IH, Keymeulen B, Mathieu C, Rottiers R, Weets I, Vandemeulebroucke E, Truyen I, Kaufman L, Schuit FC, Pipeleers DG, Gorus FK; Belgian Diabetes Registry. IA-2 autoantibodies predict impending type I diabetes in siblings of patients. Diabetologia. 2002 Dec;45(12):1658-66. doi: 10.1007/s00125-002-0949-8. Epub 2002 Nov 12. PMID 12488955
- [Derived] Vandemeulebroucke E, Keymeulen B, Decochez K, Weets I, De Block C, Fery F, Van de Velde U, Vermeulen I, De Pauw P, Mathieu C, Pipeleers DG, Gorus FK; Belgian Diabetes Registry. Hyperglycaemic clamp test for diabetes risk assessment in IA-2-antibody-positive relatives of type 1 diabetic patients. Diabetologia. 2010 Jan;53(1):36-44. doi: 10.1007/s00125-009-1569-3. Epub 2009 Nov 7. PMID 19898832